CLINICAL TRIAL: NCT05807087
Title: Prospective Randomized Study Between Conventional Techniques & Piezosurgery in the Management of Nasal Bony Pyramid
Brief Title: Comparison of Conventional Techniques & Piezosurgery in the Management of the Nasal Bony Pyramid
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hams Hamed Abdelrahman (Other)
Responsible Party: Sponsor-Investigator, Hams Hamed Abdelrahman, Assistant lecturer of DPH and Clinical statistician, Alexandria University
Organization: Alexandria University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NasalBoneSurgery_2021
Record Dates: First submitted 2023-03-15; First posted 2023-04-11 (Actual); Last update posted 2023-04-11 (Actual); Status verified 2023-03

CONDITIONS: Nasal Injury

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mechanical Osteotomy (Active Comparator)
  Interventions: Procedure: Conventional osteotomy
- Piezosurgery (Experimental)
  Interventions: Procedure: Piezosurgery osteotomy

INTERVENTIONS:
Procedure: Conventional osteotomy — The nasal skeleton was accessed using a closed approach or an open approach is done via a transcolumellar and infracartilaginous incision. Osteotomy was made using osteotomes.
  Arms: Mechanical Osteotomy
Procedure: Piezosurgery osteotomy — full exposure of the nasal bony pyramid is needed.
  Arms: Piezosurgery

SUMMARY:
It is well-known and universally acknowledged that rhinoplasty is the most demanding procedure in facial aesthetic surgery. Postoperatively nasal osteotomies result in variable degrees of edema and ecchymosis and surgeons have tried various techniques, instruments, and postoperative methods to diminish these uncomfortable morbidities. Piezosurgery is used nowadays to decrease the incidence of injured soft tissues and vital structures passing near the osteotomy line. Its use in rhinoplasty was advocated to prevent unwanted back fractures as well as to decrease bleeding while keeping the nasal mucosa intact thus minimizing postoperative sequelae.

ELIGIBILITY:
Inclusion Criteria:

* Patients requesting aesthetic rhinoplasty, post-traumatic rhinoplasty, and post-cleft nose rhinoplasty.

Exclusion Criteria:

* Patients with severe systemic disease (American Society of Anesthesiologists physical status classification system III & IV).
* Psychological disorders.
* Female patients younger than 16 years of age and male patients younger than 18 years of age.
* Patients with autoimmune and skin diseases.

Ages: 16 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 24 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2022-09-16 (Actual); Study Completion 2022-09-16 (Actual)

PRIMARY OUTCOMES:
Operative time | During procedure
  Operation duration will be calculated
Visual analogue score | immediately after procedure
  The VAS consists of a 10cm line, with two end points representing 0 ('no pain') and 10 ('pain as bad as it could possibly be')
Change in periorbital edema | Baseline and 1 week
  Grade 1 - No coverage of iris with eyelids, Grade 2 - Slight coverage of iris with swollen eyelids, Grade 3 - Full coverage of iris with swollen eyelids, Grade 4 - Full closure of eyes.
Change in eccyhmosis | Baseline and 1 week
  Grade 1 - Eccyhmosis upto the medial one-third part of lower and /or upper eyelid, Grade 2 - Ecchymosis upto the medial two-third part of the lower and/or upper eyelid. Grade 3 - Ecchymosis up to the full length and /or upper eyelid.

SECONDARY OUTCOMES:
Functional - aesthetic outcome | immediately after procedure
  The SCHNOS is a 10-item self-rated questionnaire that uses a Likert-like 0-5 scale ('no problem' to 'extreme problem'). The SCHNOS does not produce a combined total score, but two scores - one for each domain, an obstruction score (SCHNOS-O) and a cosmesis score (SCHNOS-C) The SCHNOS-O is calculated as a sum of scores of items 1-4 divided by 20 and multiplied by 100. The SCHNOS-C score is calculated as a sum of scores of items 5-10 divided by 30 and multiplied by 100.

CONTACTS AND LOCATIONS:
Locations (1):
- Outpatient Clinic of Oral and Maxillofacial Surgery Department, Faculty of Dentistry, Alexandria University, Egypt, Alexandria, Azarita, Egypt